CLINICAL TRIAL: NCT07165535
Title: Quality of Life and Care Organization of Patients With Chronic Myeloid Leukemia in the Lombardy Hematology Network
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: CML-OPERAP
Record Dates: First submitted 2025-07-28; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chronic Myeloid Leukemia (CML)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to assess the impact of the organizational model of the hematology center on the quality of life of patients with CML estimated through standardized tools (EORTC QLQ-30, CML24) and through the patient's opinion regarding aspects of the quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older.
* Subjects diagnosed with Chronic Myeloid Leukemia.
* Subjects diagnosed with CML under care at the hematology outpatient clinics of the 21 REL centers.
* Subjects followed at the reference hematology center for a minimum of 6 months.
* Freely given informed consent obtained before the start of the study.

Exclusion Criteria:

* Subjects who have not given consent to participate in the study.
* Subjects who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with Chronic Myeloid Leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-05-17 (Estimated); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Assessed Through Standardized Questionnaires (EORTC QLQ-C30) | One-time measurement at baseline during the 12-month enrollment period
  Quality of life in CML patients will be assessed using the validated EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30).
  This instrument evaluates multiple domains of physical, emotional, and social functioning, as well as general cancer-related symptoms. The questionnaire consists of 30 items, with 28 items scored from 1 (minimum functioning/symptom presence) to 4 (maximum functioning/symptom presence), and 2 items scored from 1 to 7. Raw scores are transformed according to EORTC guidelines onto a standardized scale from 0 to 100, where 0 represents the lowest functioning or symptom level and 100 represents the highest functioning or symptom level. For functional scales and the global health status, higher scores indicate better quality of life, whereas for symptom scales, higher scores indicate worse quality of life.
Quality of Life Assessed Through Standardized Questionnaires (EORTC QLQ-CML24) | One-time measurement at baseline during the 12-month enrollment period.
  Quality of life in CML patients will also be assessed using the validated EORTC QLQ-CML24 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Chronic Myeloid Leukemia 24), which measures symptoms and functioning specifically related to CML. This questionnaire includes 24 items scored from 1 to 4. Raw scores are transformed according to EORTC guidelines onto a standardized 0 to 100 scale, with 0 indicating the lowest and 100 the highest level of functioning or symptom presence. Higher scores on functional scales correspond to better quality of life, while higher scores on symptom scales correspond to worse quality of life.

SECONDARY OUTCOMES:
Evaluation of Different Organizational and Care Models of Hematology Outpatient Clinics for CML Patients | One-time measurement at baseline during the 12-month enrollment period.
  Assessment of how different organizational models of hematology outpatient clinics (e.g., structure, workflow, resource allocation) influence the patient experience and perceived quality of care within the REL network.
  Data for these outcomes will be collected through study-specific questionnaires administered to patients.
Evaluation of Strengths and Weaknesses of Different Outpatient Organizational Settings | One-time measurement at baseline during the 12-month enrollment period.
  Comparison of perceived strengths and weaknesses of various organizational settings, such as large vs. small centers and dedicated outpatient clinics vs. time-slot-based care.
  Data for these outcomes will be collected through study-specific questionnaires administered to patients.
Evaluation of Factors Affecting Daily Life in CML Patients | One-time measurement at baseline during the 12-month enrollment period.
  Assessment of the impact of CML and its management on daily living activities, autonomy, and social participation, as reported by patients.
  Data for these outcomes will be collected through study-specific questionnaires administered to patients.
Evaluation of Emotional Well-being in CML Patients | One-time measurement at baseline during the 12-month enrollment period.
  Assessment of the emotional and psychological status of patients using validated tools (e.g., emotional functioning domain of EORTC QLQ-C30).
  Data for these outcomes will be collected through study-specific questionnaires administered to patients.
Impact of CML on Family and Work Relationships | One-time measurement at baseline during the 12-month enrollment period
  Evaluation of how CML affects patients' family dynamics and work life, including ability to work, interpersonal relationships, and role functioning.
  Data for these outcomes will be collected through study-specific questionnaires administered to patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, MB, Italy